CLINICAL TRIAL: NCT02456363
Title: Anti-Tumor Necrosis Factor Therapy In Patients With Ankylosing Spondylitis-A Registry Project
Brief Title: Anti-Tumor Necrosis Factor Therapy In Patients With Ankylosing Spondylitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, GCRC, Chief, Department of Critical Care Medicine and Division of Pulmonary Medicine, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS09128
Record Dates: First submitted 2014-12-14; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Ankylosing Spondylitis
Keywords: Adalimumab; NSAIDs; safety; efficacy
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Tumor Necrosis Factors; Adalimumab; Etanercept; golimumab; Anti-Inflammatory Agents, Non-Steroidal; Sulfasalazine; Etoricoxib; Celecoxib; Meloxicam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- NSAIDs(+) and sulfasalazine(+) (Experimental): use TNF alpha: Adalimumab (Humira)、Etanercept (Enbrel) or Golimumab (Simponi) combine with use of NSAIDs and no sulfasalazine
  Interventions: Biological: TNF alpha; Drug: NSAIDs and sulfasalazine
- NSAIDs(+) and sulfasalazine(-) (Experimental): use TNF alpha: Adalimumab (Humira)、Etanercept (Enbrel) or Golimumab (Simponi) combine with use of NSAIDs and no sulfasalazine
  Interventions: Biological: TNF alpha; Drug: NSAIDs and sulfasalazine
- NSAIDs(-) and sulfasalazine(+) (Experimental): use TNF alpha: Adalimumab (Humira)、Etanercept (Enbrel) or Golimumab (Simponi) combine with use of sulfasalazine and no NSAIDs
  Interventions: Biological: TNF alpha; Drug: NSAIDs and sulfasalazine
- NSAIDs(-) and sulfasalazine(-) (Experimental): use TNF alpha: Adalimumab (Humira)、Etanercept (Enbrel) or Golimumab (Simponi) neither NSAIDs nor sulfasalazine
  Interventions: Biological: TNF alpha

INTERVENTIONS:
Biological: TNF alpha — Depending on patient need to use different TNF alpha
  Other Names: Drug: Adalimumab (Humira); Drug: Etanercept (Enbrel); Drug: Golimumab (Simponi)
Drug: NSAIDs and sulfasalazine — randomized case, combine with use of NSAIDs(-/+) and sulfasalazine(-/+)
  Other Names: Drug: Arcoxia; Drug: Celebrex; Drug: Tonec; Drug: Mobic; Drug: sulfasalazine
  Arms: NSAIDs(+) and sulfasalazine(+); NSAIDs(+) and sulfasalazine(-); NSAIDs(-) and sulfasalazine(+)

SUMMARY:
Assessed using (1) Adalimumab(Humira) and NSAIDs (2) Use only Adalimumab(Humira) treatment of ankylosing spondylitis patient safety and efficacy.

DETAILED DESCRIPTION:
In this study, single center, treatment, open, randomized, controlled clinical trial to assess Adalimumab(Humira) style with NSAIDs for the treatment of patients with ankylosing spondylitis, a total of 300 are expected to be included in the consent form signed by the subject, will be randomly assigned to treatment groups with a control group of 150 people.

Subjects to be returned in the first week outpatient follow 0,8,20,44,68,92 accept routine physical examination (weight, blood pressure, etc.), AS Scale (BASDAI, BASFI, BAS-G), fingertip ground tests, lumbar range of motion, chest expansion test, lateral bending test, the occipital bone measurements, physician global assessment (Physician global assessment), patient pain scores (VAS), AS quality of Life scale (ASQOL), SF-36 quality of life scale, Complete joint assessment, ASAS20 response criteria, assessment of laboratory analysis inflammation index (HS-CRP, IgA, ESR), safety index checks (CBC, SGPT, Serum creatinine, HBV-DNA if HbsAg (+), HCV -RNA if HCVAB.

Subjects need to return OPD week 0, accept Anti-HBs, Anti-HBc, HBsAg, Anti-HCV. Subjects required to return to the first outpatient follow 0,20,92 weeks, pulmonary function tests.

Therefore, the subjects in the 92 weeks of the trial, a total need for blood six times, each time for blood about 10 cc. And to assess side effects and adverse events (Adverse Event, AE), serious adverse events (Serious Adverse Event, SAE)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* HLA B27 positive
* X ray examination
* Clinical symptoms and physical examination, the following three conditions are subject to at least two:

  i.lower back pain and morning stiffness symptoms persist more than 3 months ii. lumbar activity is restricted iii. chest expansion is restricted
* Active disease for four weeks or more (continue two examination BASDAI>6, ESR> 28 mm/1 hr and CRP>1 mg/dl)

Exclusion Criteria:

* pregnant or breast-feeding women
* patients with active infections
* highly infectious patients
* Cancer or precancerous condition of the patient
* multiple sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-11; Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
mSASSS (Modified Stoke Ankylosing Spondylitis Spinal Score) | weeks 92
  weeks 92 of the spinal injury

CONTACTS AND LOCATIONS:
Overall Officials: Wei C- C, M.D., Study Director — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan